CLINICAL TRIAL: NCT03450408
Title: Foley Bulb Insertion by Blind Placement Versus Direct Visualization: A Randomized Controlled Trial
Brief Title: Foley Bulb Insertion Method: Blind vs. Direct
Acronym: FrIENDly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17-0359
Record Dates: First submitted 2018-02-06; First posted 2018-03-01 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The individual or individuals responsible for assessing outcome data will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placement with gloved hand (Active Comparator): The Foley bulb transcervical dilator will be placed blindly with a gloved hand.
  Interventions: Procedure: Method of placement of Foley bulb transcervical dilator
- Placement with sterile speculum (Active Comparator): The cervix will be directly visualized using a sterile speculum, and an instrument will be used to advance the Foley bulb transcervical dilator into the cervical os.
  Interventions: Procedure: Method of placement of Foley bulb transcervical dilator

INTERVENTIONS:
Procedure: Method of placement of Foley bulb transcervical dilator — This trial will assess two methods used to place a Foley bulb transcervical dilator.

SUMMARY:
The investigators will compare, in a randomized clinical trial, two methods of placement (placement with a gloved hand vs. placement with a sterile speculum) of a Foley bulb transcervical dilator. The primary outcome is rate of infection.

DETAILED DESCRIPTION:
The target population for this study is women who present for scheduled induction of labor. If there is a decision by the obstetric team to place a transcervical Foley dilator for cervical ripen-ning, the obstetric team will notify the research team so that the patient may be screened for the study. If the patient consents to participation, written informed consent will be obtained by person-to-person contact. The PI, study coordinator, or a collaborator will be responsible for the in-formed consent. After informed consent is obtained, the patient will be randomized to the study group (digital placement) or the control group (placement with a sterile speculum).

The control group will undergo induction of labor by placement via sterile speculum of a 22-French transcervical Foley catheter. The cervix is visualized with a sterile vaginal speculum and cleaned with iodine or chlorhexidine. A Foley catheter is introduced into the cervix and the bal-loon is filled with 60 ml of sterile 0.9% NaCl. The Foley catheter will be left in place for at least 12 hours, and no longer than 24 hours. After placement standard intrapartum management of the patient will ensue.

The study group will undergo induction of labor by digital blind placement of a 22-French trans-cervical Foley catheter. A Foley catheter is introduced into the cervix using digits and hands wearing sterile gloves and the balloon is filled with 60 ml of sterile 0.9% NaCl. The Foley catheter will be left in place for at least 12 hours, and no longer than 24 hours. After placement standard intrapartum management of the patient will ensue.

If cervix remains unfavorable after extraction of the dilators (< 3cm and at most 60% effaced), a second Foley catheter will be used in this case for a maximum of 12 hrs. No crossover will be allowed. In other words, a second Foley bulb will be placed in the same manner as the first assignment arm.

In any attempts, if the Foley bulb is not able to be placed in either insertion technique , a prostaglandin agent for cervical ripening may be used and insertion of the mechanical dilator can be re-attempted at a later time, as is the standard of care at our institution. No cross over will be allowed.

This will be an unblinded randomized clinical trial.

No significant adverse effects are expected with the use of transcervical Foley catheters for mechanical dilation. The most significant risks are vaginal bleeding due to cervical trauma and incidental rupture of membranes, as well as pain or discomfort with placement. The patient will undergo inpatient induction of labor, so any adverse reaction would be promptly detected and addressed.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 50 years
* Induction of labor
* Plan for Foley bulb placement by the managing obstetrics team

Exclusion Criteria:

* Patient unwilling or unable to provide consent
* Fetal demise or major congenital anomaly
* Immunosuppressed patients: i.e., taking systemic immunosuppressants or steroids (e.g. transplant patients; not including steroids for lung maturity), HIV with CD4<200, or other
* Fever (>38°C) in the 48 hours prior to presentation for induction of labor
* Use of anti-pyretic agent (i.e., acetaminophen) in the eight hours preceding admission for induction of labor

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — As we are assessing pregnant patients, participants will be female.
Enrollment: 372 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Infection | Labor to 30 days postpartum
  Pooled maternal infection

SECONDARY OUTCOMES:
Maternal fever | From beginning of labor process to time of discharge, up to seven days
  Greater than or equal to 38 degrees Celsius
Request for pain relief | Within 30 minutes of placement procedure
  Request for IV pain medications or epidural placement
Vaginal bleeding | Within 30 minutes of placement procedure
  In the time period immediately following placement
Artificial rupture of membranes | At time of placement of Foley bulb transcervical dilator
  Rupture of amniotic sac
Chorioamnionitis or "triple I" | From beginning of labor process until time of delivery
  Presumptive or confirmed diagnosis
Endometritis | From time of delivery to 30 days postpartum
  Postpartum intrauterine infection

CONTACTS AND LOCATIONS:
Overall Officials: Antonio F Saad, MD, Study Chair — University of Texas
Locations (1):
- University of Texas Medical Branch John Sealy Hospital, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kuhlmann MJ, Spencer N, Garcia-Jasso C, Singh P, Abdelwahab M, Vaughn M, Marshall K, Prasad N, Soulsby-Monroy R, Saade GR, Saad AF. Foley Bulb Insertion by Blind Placement Compared With Direct Visualization: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jan 1;137(1):139-145. doi: 10.1097/AOG.0000000000004182. PMID 33278290